CLINICAL TRIAL: NCT04223362
Title: PICk-UP: PersonalIsed CommUnity-based Physical Activities for Patients With Chronic Obstructive Pulmonary Disease
Acronym: PICk UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Câmara Municipal de Aveiro (Unknown); Câmara Municipal de Estarreja (Unknown); Centro Hospitalar do Baixo Vouga (Other); Administração Regional de Saúde do Centro (Other); Escola Superior de Saúde da Universidade de Aveiro (Unknown); Instituto de Biomedicina da Universidade de Aveiro (Unknown)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Associate Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFRH/BD/148738/2019
Record Dates: First submitted 2019-12-19; First posted 2020-01-10 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: COPD
Keywords: Physical activity; Community; Behavioural change; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blind, outcome assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary rehabilitation + Community-based physical activity programme (Experimental): After pulmonary rehabilitation, the experimental group will integrate a community-based physical activity programme.
  Interventions: Other: Community-based physical activity programme; Other: Pulmonary Rehabilitation
- Pulmonary Rehabilitation (Active Comparator): The control group will only receive pulmonary rehabilitation, which integrates physical activity recommendations.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Community-based physical activity programme — After completing a pulmonary rehabilitation programme, participants will enrol a 6-months personalised community-based physical activity programme, which will include 2 sessions/week, with the aerobic training being the cornerstone. Patients will receive the PICk UP manual and a diary to register their physical activities. During the 1st month the physiotherapist will guide patients through 4 types of outdoors and indoors physical activities. Patients will then be asked to choose and commit to 1 or 2 activities, according to their preferences, which they shall integrate for another 5 months. During this period, the support provided by physiotherapist will decrease over time.
  Arms: Pulmonary rehabilitation + Community-based physical activity programme
Other: Pulmonary Rehabilitation — Patients will receive the same pulmonary rehabilitation programme as the experimental group, i.e., exercise training twice a week and education and psychosocial support once every other week, which integrates physical activity recommendations.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a major individual, social and economic burden worldwide. Pulmonary rehabilitation is a fundamental evidence-based intervention to manage COPD. However, pulmonary rehabilitation benefits tend to decline over time and sustaining a long-term physical activity lifestyle is challenging, leading to worse health-related quality of life. Personalised post-pulmonary rehabilitation programmes, combining different physical activities modalities with social interaction, are warranted to enable a shift from a disease-based to a patient-centred model and encourage a sustainable behavioural change. Although such programmes have the potential to sustain pulmonary rehabilitation benefits and promote patients' long-term adherence to physical activity, their availability within the community is scarce. Hence, the investigators will implement a personalised community-based physical activity programme (PICk UP), using the available resources, adapted to patient's needs/preferences. PICk UP will be a sustainable response to support healthy lifestyles and enhance pulmonary rehabilitation benefits of respiratory patients, by integrating them within the community and embracing urban facilities.

The aim of this study is to assess the effectiveness of PICk UP, a personalised community-based physical activity programme, tailored to patients' needs and preferences, on their physical activity levels.

It is expected that PICk UP will empower patients to remain physically active and foster the maintenance of pulmonary rehabilitation benefits.

DETAILED DESCRIPTION:
COPD-related morbidity and mortality has been increasing, making COPD already the third leading cause of death and a growing global health concern.

Pulmonary rehabilitation (PR) is a comprehensive intervention, with known cost-effectiveness in managing patients with COPD. One of the PR goals is to improve physical activity (PA), since it has shown to reduce exacerbations and mortality.

Nevertheless, adopting/sustaining a physically active behaviour is highly challenging and benefits of PR are usually lost 6 months after its completion. Therefore, PA programmes capable to maintain the PR effects are urgently needed Community can provide different PA modalities in various settings, which can be personalised to patients' needs and preferences. By filling the gaps between healthcare systems and patients' daily environment, these programmes have the potential to improve patients' HRQoL and self-efficacy, enhancing their ability to overcome exercise barriers and their motivation to sustain a physically active behaviour.

PICk UP will offer patients different PA modalities tailored to their preferences and needs, thus personalising the community programmes, and aiming at sustaining a physically active behaviour and enhancing their HRQoL.

This study aims at assessing the effectiveness of PICk UP, a personalised community-based physical activity programme tailored to patients' needs and preferences, on their physical activity levels and on the maintenance of pulmonary rehabilitation benefits. To accomplish these aims a randomised controlled trial will be conducted.

PICk UP randomised controlled trial

The primary aim of this study is to assess the effectiveness of PICk UP, a personalised community-based PA programme, tailored to patients' needs and preferences, on their PA levels.

The secondary aims is to determine the short- and mid-term effects of PICk UP on HRQoL symptoms, number of exacerbations, healthcare use, exercise capacity, functionality, motivation to exercise, peripheral muscle strength and emotional status.

Recruitment Primary healthcare providers of Aveiro and Estarreja or pulmonologists of the Centro Hospitalar do Baixo Vouga will inform eligible patients about the study. Additional information will be provided to those interested to participate in a meeting with the researcher and written informed consent will be acquired. Patients with COPD will be eligible if they are clinically stable, as determined by their referred doctor, and completed a PR programme in the previous month. Patients will be excluded if they present signs of cognitive impairment or have significant cardiovascular, neurological or musculoskeletal diseases, which may limit their participation.

Study design Patients will be randomised into experimental group (EG) or control group (CG). The EG will receive the PICk UP programme. The CG will receive no additional interventions and will only proceed with the physical activity recommendations delivered during the pulmonary rehabilitation programme. Assessments will be conducted by a second researcher blinded to the intervention.

Data collection:

Data will be collected at baseline, after 3 months and after the intervention (6 months). The researcher will collect:

* Sociodemographic, anthropometric, general clinical data (e.g., number of exacerbations or healthcare utilisation);
* Physical activity levels (time in sedentary, moderate and vigorous physical activities; steps/day): accelerometry.
* Health related quality of life: St. George's Respiratory Questionnaire.
* Disease impact: COPD Assessment Test.
* Exercise tolerance: six-minute walk test.
* Motivations to exercise: Behavioural Regulation and Exercise Questionnaire-3.
* Quadriceps muscle strength: Handheld dynamometry.
* Fatigue: Checklist of Individual Strength-8 and the Functional assessment of chronic illness therapy fatigue subscale;
* Handgrip strength: dynamometry.
* Emotional status: Hospital Anxiety and Depression Scale.
* Occurrence of adverse events and adherence to the interventions

Intervention:

Participants in the EG will enrol a 6-months personalised community-based physical activity programme, which will include 2 sessions/week, with the aerobic training being the cornerstone. Patients will receive the PICk UP manual and a diary to register their physical activities. During the 1st month the physiotherapist will guide patients through 4 types of outdoors (e.g., walking, cycling trails) and indoors (e.g., dance, pilates) physical activities. Patients will then be asked to choose and commit to 1 or 2 activities, according to their preferences, which they shall integrate for another 5 months. During this period, the support provided by physiotherapist will decrease over time

* 2nd and 3rd months: support every 2-weeks (face-to-face physical activity sessions alternated with phone-calls) to reassure safety, clarify doubts, monitor patients' evolution and enhance their motivation to physical activity;
* 4th month: 1 face-to-face physical activity session;
* 5th month: 1 phone-call;
* 6th month: no support. The sport-related professionals will register patients' attendance to the programme.

Sample size estimation:

The sample size was estimated using G*Power 3.1.9.6, with an effect size specification "as in G*Power 3.0", for the within-between interaction of a repeated measures ANOVA with two groups (control and experimental) and 3 measurements (immediately after, 3 and 6 months post-PR) of the defined primary outcome (time in moderate to vigorous PA). The investigators considered an α of 0.05, a power of 0.80, a repeated measures correlation of 0.5, a nonsphericity correction of 1 and an expected effect size f of 0.30. The effect size f was derived from the partial η2 of 0.21 (f=0.516) obtained from a study which aimed to assess the impact of a PA-focused behavioural intervention during and after PR on PA levels in patients with COPD. A smaller f value of 0.30 was chosen to account for a longer follow-up period (up to 6 months after PR, instead of 3) and differences in selected time-points. The calculated sample size was 20 (i.e., 10 in each group) COPD patients and considering a possible 50% dropout rate, the final sample size was determined to be 40.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of a chronic obstructive pulmonary disease
* clinically stable in the previous month (no changes in medication or occurrence of acute exacerbations)
* ≥ 18 years old
* able to provide their own informed consent
* patients classified as a GOLD C or D (according to the global initiative for chronic obstructive pulmonary disease criteria), or classified as GOLD B and present a FEV1%predicted<30%, or present peripheral oxygen saturation ≤90% at rest or <85 during the 6MWT must be previously assessed by pneumologist or physiatrist.

Exclusion Criteria:

* Signs of cognitive impairment;
* Neoplasic /immunologic disease or an unstable/significant cardiac, musculoskeletal, neuromuscular or psychiatric condition limiting the ability to exercise or co-operate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in physical activity levels (time spent in moderate to vigorous physical activities) | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Accelerometer-based activity monitors. Time spent in moderate and vigorous physical activities during the day, will be collected with the activity monitors GT3X+ (ActiGraph) during one week.

SECONDARY OUTCOMES:
Change in time spent in sedentary physical activities | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Accelerometer-based activity monitors. Time spent in sedentary physical activities during the day, will be collected with the activity monitors GT3X+ (ActiGraph) during one week.
Change in steps per day | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Accelerometer-based activity monitors. Number of steps/day will be collected with the activity monitors GT3X+ (ActiGraph) during one week.
Change in Health-related quality of life - St. George Respiratory Questionnaire. | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  St. George Respiratory Questionnaire (SGRQ) will be used to assess Health Related quality-of-life. The SGRQ is a comprehensive well-established 50-item questionnaire to measure health status in patients with COPD. Scores can be provided for each domain (symptoms, activities and impact) and as a total score, ranging from 0 (no impairment) to 100 (worst possible health status).
Change in exercise tolerance - 6MWT | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Exercise capacity will be tested in a 6-minute walk test, since it allows exercise prescription. The test results will be presented as the walked distance (meters).
Change in quadriceps muscle strength | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Quadriceps muscle strength will be measured using a handheld dynamometer (kilogram/force).
Change in overall functionality - physical performance test | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Functionality will be tested with the physical performance test (PPT), which assesses multiple domains of physical function using tasks that simulate activities of daily living. This measure has 9-items with a total score of 36 points, with higher scores indicating better performance.
Change in frequency of exacerbations | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Number of exacerbations in the previous year, which are related to COPD decline
Change in handgrip strength | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  handgrip strength will be measured with a dynamometer (kg)
Change in motivation to exercise - Behavioutal regulation exercise scale | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  The Behavioural Regulation Exercise Scale-3 (BREQ-3) will be used to assess behavioural regulation under the self-determination theory in the exercise domain. The BREQ-3 has 24 itens with a 5-point Likert scale grouped into 6 factors (ammotivation, external regulation, introjected regulation, identified regulation, integrated regulation and intrinsic motivation). Those represent different forms of regulation, going from non-self determined to completely self-determined regulation. Scores per subscale range from 0 (not true to the participant) to 4 (very true to the participant), with higher scores indicating a better result.
Change in Physical activity | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  The Brief Physical Activity questionnaire will be used to assess physical activity. It a 2 items questionnaire, with scores ranging from 0 to 8 and higher scores representing better results. If the sum of the two items score is above or equal 4 the subject will be considered physically active.
Change in symptom's impact in patients' life | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  COPD Assessment Test (CAT) will be used to assess burdensome symptoms in patients' life with 8 items (cough, sputum, dyspnoea, chest tightness, capacity of exercise and home daily activities, confidence leaving home, sleep and energy levels). The scores range from 0-40, organised in 4 categories, namely <10 low impact, 10-20 medium, 21-30 high and >30 very high impact, with 5 representing the upper limit of normal in healthy non-smokers
Change in Emotional state | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Hospital Anxiety and Depression Scale will be used to assess symptoms of anxiety and depression. It is a 14 item questionnaire that can be subdivided in two subscales: anxiety and depression. Scores are provided for each subscale and range from 0 to 21, with higher scores meaning more symptoms of anxiety and depression.
Change in experience of fatigue | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  The fatigue subscale of the Checklist of Individual Strength (CIS-FS) will be used to assess fatigue. The subscale is an 8-item questionnaire, with higher scores indicating higher levels of fatigue. The total scores range from 8 to 56.
Change in impact and experience of fatigue | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  The Functional assessment of cancer therapy - fatigue subscale will be used to assess fatigue levels. It is multi-dimensional 13-item questionnaire assessing tiredness, weakness and difficulty in handling daily activities due to fatigue. Scores range from 0 to 52, with higher scores indicating less fatigue.
Change in Healthcare utilization (number of participants visiting emergency department) | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Healthcare utilization will be assessed through the number of participants that visit emergency department.
Change in Healthcare utilization (number of visits of each participant to the emergency department) | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Healthcare utilization will be assessed through the number of visits of each participant to the emergency department in the previous year.
Change in Healthcare utilization (number of hospital admissions) | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Healthcare utilization will be assessed through the number of hospital admissions each participant had in the previous year.
Change in Healthcare utilization (duration of hospital admissions) | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Healthcare utilization will be assessed through the duration (in days) of hospital admissions each participant had in the previous year.
Adherence to the PICk UP programme | Adherence will be collected in each session of physical activity throughout the 6 months.
  Participants' from the EG adherence to the physical activity programme will be registered by the sports professional responsible for each physical activity and also by participants' using a diary.
Occurrence of adverse events | Occurrence of an adverse event will be collected in each session of physical activity throughout the 6 months.
  The occurrence of adverse events in participants from the EG during the PICk UP programme will be registered by the sports professional responsible for each physical activity and also by participants' in their diaries.

OTHER OUTCOMES:
Change in Body Mass Index | Multiple time points through study completion - immediately after pulmonary rehabilitation and up to 3 and 6 months after pulmonary rehabilitation.
  Patients' body mass index will be assessed in kg/m^2 based on patients' height and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Alda S. Marques, Principal Investigator — : School of Health Sciences of the University of Aveiro (ESSUA)
Locations (1):
- University of Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gimeno-Santos E, Frei A, Steurer-Stey C, de Batlle J, Rabinovich RA, Raste Y, Hopkinson NS, Polkey MI, van Remoortel H, Troosters T, Kulich K, Karlsson N, Puhan MA, Garcia-Aymerich J; PROactive consortium. Determinants and outcomes of physical activity in patients with COPD: a systematic review. Thorax. 2014 Aug;69(8):731-9. doi: 10.1136/thoraxjnl-2013-204763. Epub 2014 Feb 20. PMID 24558112
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Beauchamp MK, Evans R, Janaudis-Ferreira T, Goldstein RS, Brooks D. Systematic review of supervised exercise programs after pulmonary rehabilitation in individuals with COPD. Chest. 2013 Oct;144(4):1124-1133. doi: 10.1378/chest.12-2421. PMID 23429931
- [Background] Jenkins AR, Gowler H, Curtis F, Holden NS, Bridle C, Jones AW. Efficacy of supervised maintenance exercise following pulmonary rehabilitation on health care use: a systematic review and meta-analysis. Int J Chron Obstruct Pulmon Dis. 2018 Jan 10;13:257-273. doi: 10.2147/COPD.S150650. eCollection 2018. PMID 29391784
- [Background] Rochester CL, Spruit MA. Maintaining the Benefits of Pulmonary Rehabilitation. The Holy Grail. Am J Respir Crit Care Med. 2017 Mar 1;195(5):548-551. doi: 10.1164/rccm.201609-1925ED. No abstract available. PMID 28248138
- [Background] McNamara RJ, McKeough ZJ, Mo LR, Dallimore JT, Dennis SM. Community-based exercise training for people with chronic respiratory and chronic cardiac disease: a mixed-methods evaluation. Int J Chron Obstruct Pulmon Dis. 2016 Nov 16;11:2839-2850. doi: 10.2147/COPD.S118724. eCollection 2016. PMID 27895476
- [Background] Robinson H, Williams V, Curtis F, Bridle C, Jones AW. Facilitators and barriers to physical activity following pulmonary rehabilitation in COPD: a systematic review of qualitative studies. NPJ Prim Care Respir Med. 2018 Jun 4;28(1):19. doi: 10.1038/s41533-018-0085-7. PMID 29867117
- [Background] Desveaux L, Harrison S, Lee A, Mathur S, Goldstein R, Brooks D. "We are all there for the same purpose": Support for an integrated community exercise program for older adults with HF and COPD. Heart Lung. 2017 Jul-Aug;46(4):308-312. doi: 10.1016/j.hrtlng.2017.04.008. Epub 2017 May 17. PMID 28527832
- [Background] Cecins N, Landers H, Jenkins S. Community-based pulmonary rehabilitation in a non-healthcare facility is feasible and effective. Chron Respir Dis. 2017 Feb;14(1):3-10. doi: 10.1177/1479972316654287. Epub 2016 Jul 8. PMID 27315829
- [Background] Breda J, Jakovljevic J, Rathmes G, Mendes R, Fontaine O, Hollmann S, Rutten A, Gelius P, Kahlmeier S, Galea G. Promoting health-enhancing physical activity in Europe: Current state of surveillance, policy development and implementation. Health Policy. 2018 May;122(5):519-527. doi: 10.1016/j.healthpol.2018.01.015. Epub 2018 Feb 3. PMID 29422372
- [Background] Rabinovich RA, Louvaris Z, Raste Y, Langer D, Van Remoortel H, Giavedoni S, Burtin C, Regueiro EM, Vogiatzis I, Hopkinson NS, Polkey MI, Wilson FJ, Macnee W, Westerterp KR, Troosters T; PROactive Consortium. Validity of physical activity monitors during daily life in patients with COPD. Eur Respir J. 2013 Nov;42(5):1205-15. doi: 10.1183/09031936.00134312. Epub 2013 Feb 8. PMID 23397303
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] O'Shea SD, Taylor NF, Paratz JD. Measuring muscle strength for people with chronic obstructive pulmonary disease: retest reliability of hand-held dynamometry. Arch Phys Med Rehabil. 2007 Jan;88(1):32-6. doi: 10.1016/j.apmr.2006.10.002. PMID 17207672
- [Background] Cid L, Monteiro D, Teixeira D, Teques P, Alves S, Moutao J, Silva M, Palmeira A. The Behavioral Regulation in Exercise Questionnaire (BREQ-3) Portuguese-Version: Evidence of Reliability, Validity and Invariance Across Gender. Front Psychol. 2018 Oct 11;9:1940. doi: 10.3389/fpsyg.2018.01940. eCollection 2018. PMID 30364299
- [Background] Polkey MI, Qiu ZH, Zhou L, Zhu MD, Wu YX, Chen YY, Ye SP, He YS, Jiang M, He BT, Mehta B, Zhong NS, Luo YM. Tai Chi and Pulmonary Rehabilitation Compared for Treatment-Naive Patients With COPD: A Randomized Controlled Trial. Chest. 2018 May;153(5):1116-1124. doi: 10.1016/j.chest.2018.01.053. Epub 2018 Apr 3. PMID 29625777
- [Background] Marques A, Jacome C, Cruz J, Gabriel R, Brooks D, Figueiredo D. Family-based psychosocial support and education as part of pulmonary rehabilitation in COPD: a randomized controlled trial. Chest. 2015 Mar;147(3):662-672. doi: 10.1378/chest.14-1488. PMID 25340477
- [Background] Fischer MJ, Scharloo M, Abbink JJ, van 't Hul AJ, van Ranst D, Rudolphus A, Weinman J, Rabe KF, Kaptein AA. Drop-out and attendance in pulmonary rehabilitation: the role of clinical and psychosocial variables. Respir Med. 2009 Oct;103(10):1564-71. doi: 10.1016/j.rmed.2008.11.020. Epub 2009 May 29. PMID 19481919
- [Background] Marques A, Jacome C, Rebelo P, Paixao C, Oliveira A, Cruz J, Freitas C, Rua M, Loureiro H, Peguinho C, Marques F, Simoes A, Santos M, Martins P, Andre A, De Francesco S, Martins V, Brooks D, Simao P. Improving access to community-based pulmonary rehabilitation: 3R protocol for real-world settings with cost-benefit analysis. BMC Public Health. 2019 May 31;19(1):676. doi: 10.1186/s12889-019-7045-1. PMID 31151409
- [Background] Webster K, Cella D, Yost K. The Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System: properties, applications, and interpretation. Health Qual Life Outcomes. 2003 Dec 16;1:79. doi: 10.1186/1477-7525-1-79. PMID 14678568
- [Background] Vercoulen JH, Swanink CM, Fennis JF, Galama JM, van der Meer JW, Bleijenberg G. Dimensional assessment of chronic fatigue syndrome. J Psychosom Res. 1994 Jul;38(5):383-92. doi: 10.1016/0022-3999(94)90099-x. PMID 7965927
- See also: Global Initiative for Chronic Obstructive Lung Disease. Global Strategy for Diagnosis, Management, and Prevention of Chronic Obstructive Pulmonary Disease 2020 report. The Global Initiative for Chronic Obstructive Lung Disease, Inc. 2020. — https://goldcopd.org/wp-content/uploads/2019/11/GOLD-2020-REPORT-ver1.0wms.pdf